CLINICAL TRIAL: NCT00132626
Title: Dynamic SPECT Imaging With [123I]ß-CIT in Patients With Parkinsonism
Brief Title: Study of Brain Imaging With Nuclear Technology in Individuals With Parkinsonian Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Molecular NeuroImaging (Other); National Institutes of Health (NIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dopamine Transporter Imaging
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Parkinson's Disease; Parkinsonian Syndrome
Keywords: parkinson; diagnosis
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Disease

INTERVENTIONS:
Drug: [123I]ß-CIT and SPECT imaging

SUMMARY:
This study assesses dopamine transporter density using single photon emission computed tomography (SPECT) brain imaging with an investigational radiopharmaceutical, [123I]ß-CIT, in research participants with Parkinson's disease.

DETAILED DESCRIPTION:
The brain imaging is conducted at the Institute for Neurodegenerative Disorders in New Haven, Connecticut. The imaging procedure occurs over a two day period.

After a screening visit, including review of the potential subject's neurological history and a thorough neurologic exam, subjects are injected with [123I]ß CIT, an investigational radioactive material that localizes in the brain.

Twenty-four hours later study participants return to the Institute for Neurodegenerative Disorders where an investigational scanning procedure is used to obtain SPECT (single photon emission computed tomography) images of the brain.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Normal screening laboratory studies
* At least two of the following: resting tremor, cogwheel rigidity, bradykinesia, and postural reflex impairment

Exclusion Criteria:

* Pregnancy
* Significant medical disease including abnormalities found on screening

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1992-09; Study Completion 2005-08

PRIMARY OUTCOMES:
CIT uptake: measurement of dopamine transporter density compared with the clinical severity of illness

SECONDARY OUTCOMES:
Measurement of variability of strital uptake of [123I]ß-CIT when more than one scan has occurred

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Marek, MD, Principal Investigator — Institute for Neurodegenerative Disorders